CLINICAL TRIAL: NCT01896778
Title: Body Warming to Alter [Thermo] Regulation and the Microenvironment [B-WARM] Therapy: A Pilot Study
Brief Title: Body Warming in Improving Blood Flow and Oxygen Delivery to Tumors in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: I 229812; NCI-2013-01198 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 229812 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Adult Liver Carcinoma; Breast Carcinoma; Colon Carcinoma; Kidney Neoplasm; Lung Carcinoma; Malignant Head and Neck Neoplasm; Malignant Neoplasm; Melanoma; Ovarian Neoplasm; Soft Tissue Sarcoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Breast Neoplasms; Colonic Neoplasms; Kidney Neoplasms; Lung Neoplasms; Head and Neck Neoplasms; Neoplasms; Melanoma; Ovarian Neoplasms; Sarcoma | interventions — Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (B-WARM for 30 minutes) (Experimental): Patients undergo B-WARM at 39 degrees C for 30 minutes.
  Interventions: Procedure: Hyperthermia Treatment; Other: Laboratory Biomarker Analysis
- Arm II (B-WARM for 2 hours) (Experimental): Patients undergo B-WARM at 39 degrees C for 2 hours.
  Interventions: Procedure: Hyperthermia Treatment; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Hyperthermia Treatment — Undergo B-WARM
  Other Names: Clinical Hyperthermia; Diathermy; Hyperthermia; Hyperthermia Therapy
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized pilot clinical trial studies body warming in improving blood flow and oxygen delivery to tumors in patients with cancer. Heating tumor cells to several degrees above normal body temperature may kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and efficacy of 2 different Body Warming to Alter (Thermo) Regulation and the Microenvironment (B-WARM) regimens on altering tumor blood flow in patients with a variety of malignancies.

SECONDARY OBJECTIVES:

I. To determine if duration and thermal dose of B-WARM changes duration and extent of tumor blood flow changes in patients with a variety of malignancies.

OUTLINE: Patients are randomized to 1of 2 arms.

ARM I: Patients undergo B-WARM at 39 degrees Celsius (C) for 30 minutes.

ARM II: Patients undergo B-WARM at 39 degrees C for 2 hours.

After completion of study, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a variety of malignancies (i.e., melanoma, sarcoma, colon, head and neck, renal, breast, lung, ovary, liver)
* Patients must have measurable disease (1.0 cm or greater) by computed tomography (CT) scan
* Have an estimated glomerular filtration rate (eGFR) (using the Cockcroft-Gault equation) of more than 60 mL/min
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients of child-bearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* History of prior myocardial infarction or arrhythmia
* History of any condition deemed by the principal investigator to be a contraindication to B-WARM therapy (e.g., skin reaction, dysregulation of thermoregulation, etc)
* All patients with transdermal patches (e.g.; fentanyl, Lidoderm, scopolamine, etc)
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the patient an unsuitable candidate to receive B-WARM
* Received an investigational agent within 30 days prior to enrollment
* Received any systemic therapy within 21 days prior to planned B-WARM therapy

  * Patients may be enrolled on study but at least 21 days should elapse prior to date of B-WARM therapy
* Patients should not have either CT scanning or B-WARM if they have a fever at the time

  * Fever should be worked up and treated as appropriate
  * Patients should be afebrile for 24 hours prior to scanning or B-WARM therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-10-04 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Changes in tumor vascular (blood flow, blood volume) | Baseline to 24-88 hours
  The primary analysis will be implemented using an analysis-of-covariance model for both blood flow and blood volume.

SECONDARY OUTCOMES:
Changes in tumor vascular measures | Baseline to 88-264 hours
Incidence of adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 days post-treatment
  The frequency of toxicities will be tabulated by grade across all dose levels and cycles. The frequency of toxicities will also be tabulated for the dose estimated to be the maximum tolerated dose.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States